CLINICAL TRIAL: NCT03143036
Title: Phase 2 Study of Daratumumab in Combination With Thalidomide and Dexamethasone in Relapse and / or Refractory Myeloma
Brief Title: Daratumumab, Thalidomide and Dexamethasone in Relapse and/or Refractory Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Janssen, LP (Industry); International Myeloma Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMN004
Record Dates: First submitted 2017-04-13; First posted 2017-05-08 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-05

CONDITIONS: Relapse and / or Refractory Myeloma
Keywords: daratumumab
MeSH Terms: conditions — Recurrence; Neoplasms, Plasma Cell | interventions — daratumumab; Thalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a phase 2 study of the combination of Daratumumab, thalidomide and dexamethasone in 100 Asian patients with relapse or refractory multiple myeloma.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab, thalidomide and dexamethasone (Experimental)
  Interventions: Drug: Daratumumab, thalidomide and dexamethasone

INTERVENTIONS:
Drug: Daratumumab, thalidomide and dexamethasone — Patients will be treated with with the following schedule. IV daratumumab 16mg/kg body weight weekly for weeks 1-8 followed by daratumumab 16mg/kg body weight once every 2 weeks from weeks 9 to 24 and then daratumumab 16mg/kg once every 4 weeks from weeks 25 onwards until disease progression; PO thalidomide 100mg daily for 1 year and PO Dexamethasone 40mg (starting dose of dexamethasone is 20mg once weekly for patients >75 years old) once weekly for 1 year (13 cycles, each cycle is 4 weeks). After 1 year, patient only continue on daratumumab until progression
  Patients will be assessed every 28 days (+/-10 days).

SUMMARY:
Myeloma patients who relapse after prior treatment with bortezomib and lenalidomide have survival of less than 1 year. A number of new drugs have been approved for the treatment of relapse myeloma in the last couple of years, including, Elotuzumab, Panobinostat, Ixazomib, carfilzomib and Pomalidomide. However, most of these drugs either do not have good single agent activity or still belongs to the category of immunomodulatory drugs or proteasome inhibitors. Daratumumab is a monoclonal antibody against CD38 that is highly expressed on myeloma plasma cells. In phase ½ studies, it has impressive single agent activity in relapse and refractory myeloma with a very acceptable toxicity profile. This set the stage for combinations with daratumumab to increase efficacy and improve outcome of patients with myeloma. The use of immunomodulatory drugs, such as thalidomide and lenalidomide, has been shown to augment NK cell activity. NK cells are important mediator of antibody dependent cellular cytotoxicity. We therefore hypothesize that the combination of Daratumumab with thalidomide may therefore improve the efficacy of the treatment.

In this study, we will plan to perform a phase II trial using the Daratumumab, Thalidomide, Dexamethasone combination in 100 myeloma patients with relapse myeloma in Asia.

DETAILED DESCRIPTION:
Daratumumab is a humanized antibody against CD38 which is expressed on myeloma cells. Daratumumab exhibited single agent activity in myeloma and is a promising new treatment. Recently, 2 phase 1 / 2 studies establishes the dosing regimen for Daratumumab and impressive single agent activity of about 30% response rates in patients who relapse after prior lenalidomide and bortezomib. Daratumumab also appear to be well tolerated. The most common toxicity is infusion-related and almost all confined to the first cycle. On the whole these are manageable with early intervention, concurrent corticosteroids and anti-histamines as well as slowing infusion rate. More recently, early results from 2 randomise study comparing Daratumumab plus lenalidomide and dexamethasone compared to lenalidomide and dexamethasone, and Daratumumab plus bortezomib and dexamethasone compared to bortezomib and dexamethasone, showed that the addition of Daratumumab significantly improved response and progression free survival, including a high minimal residual disease (MRD) negative rate of more than 20% in the relapse myeloma populations.

In addition, the use of immunomodulatory drugs, such as thalidomide and lenalidomide, has been shown to augment NK cell activity. NK cells are important mediator of antibody dependent cellular cytotoxicity, which is an important mechanism of action for Daratumumab. Furthermore, in the studies using another antibody target SLAMF7, Elotuzumab, the addition of dexamethasone greatly improve efficacy. Furthermore, thalidomide plus dexamethasone combination have a long history in myeloma and is relatively well tolerated and cost-effective. We therefore propose to add Daratumumab to thalidomide and dexamethasone, as this combination will be relatively easy to deliver in the Asian population because of availability and there is good rationale that such a combination will be synergistic and well-tolerated

Patients will be assessed every 28 days (+/-10 days). Patients shall receive the treatment until disease progression, unacceptable toxicity as determined by treating physician, withdrawal of consent or mortality (whichever occurs first). After disease progression, the treating physician should provide long-term follow-up data on disease status and survival. For patients who discontinued treatment before disease progression occurred, disease assessment measurements shall be performed once every 28 days (+/- 10 days) until disease progression. After patients have documented progression of disease, they will be followed for survival every 3 months (+/-10 days) until study closure or until patients withdraws consent, is lost to follow-up or until death, whichever comes first. For any patient who is lost to follow-up, the study site shall attempt to ascertain survival information via public database search.

ELIGIBILITY:
Inclusion Criteria:

1. Multiple myeloma, diagnosed according to standard criteria, with relapsing and refractory disease at study entry
2. Patients must have evaluable multiple myeloma with at least one of the following (within 21 days of starting treatment)

   1. Serum M-protein ≥ 0.5g/dL, or
   2. In subjects without detectable serum M-protein, Urine M-protein ≥ 200mg/24 hour, or serum free light chai (sFLC) > 100mg/L (involved light chain) and an abnormal kappa/Lambda ratio
3. Must receive at least 1 line of prior treatment. (Induction therapy followed by stem cell transplantation and consolidation/maintenance therapy will be considered as one line of treatment)
4. Must have relapsed disease and/or be refractory to prior treatment except for thalidomide or lenalidomide. Refractoriness is defined as disease progression on treatment or progression within 6 months after the last dose of a given therapy. Relapse is defined according to the criteria of IMWG
5. Males and females ≥ 18 years of age or > country's legal age for adult consent
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
7. Patients must meet the following clinical laboratory criteria with 21 days of starting treatment:

   1. Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet ≥ 50,000/mm3 (≥ 30,000/mm3 if myeloma involvement in the bone marrow is >50%)
   2. Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   3. Calculated creatinine clearance ≥ 30mL/min.
8. Written informed consent in accordance with federal, local and institutional guidelines

Exclusion Criteria:

1. Female patients who are lactating or pregnant
2. Multiple Myeloma of IgM subtype
3. Glucocorticoid therapy (prednisolone > 30mg/day or equivalent) within 14 days prior to informed consent obtained
4. POEMS syndrome
5. Plasma cell leukemia or circulating plasma cells ≥ 2 x 109/L
6. Waldenstrom's Macroglobulinaemia
7. Existing peripheral neuropathy of grade 2 or higher or presence of neuropathic pain
8. Patients with known amyloidosis
9. Chemotherapy with approved or investigation anticancer therapeutics within 21 days prior to starting Dara-TD treatment
10. Focal radiation therapy within 7 days prior to start of Dara-TD. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to start of pomalidomide
11. Immunotherapy (excluding steroids) 21 days prior to start of Dara-TD
12. Major surgery (excluding kyphoplasty) within 28 days prior to start of Dara-TD
13. Active congestive heart failure (New York Heart Association [NYHA] Class III or IV), symptomatic ischaemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 4 months prior to informed consent obtained
14. Known HIV seropositive, hepatitis C infection, and/or hepatitis B (except for patients with hepatitis B surface antigen or core antibody receiving and responding to antiviral therapy directed at hepatitis B: these patients are allowed)
15. Patients with known cirrhosis
16. Patients with creatinine clearance <30m/min
17. Second malignancy within the past 3 years except:

    1. Adequately treated basal cell or squamous cell skin cancer
    2. Carcinoma in situ of the cervix
    3. Breast carcinoma in situ with full surgical resection
18. Patients with myelodysplastic syndrome
19. Patients with steroid or thalidomide hypersensitivity
20. Patients previously treated with daratumumab or other anti-CD38 antibodies.
21. Ongoing graft-versus-host disease
22. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to starting Dara-TD treatment
23. Disease refractory to thalidomide or lenalidomide
24. Contraindication to any of the required concomitant drugs or supportive treatments
25. Any clinically significant medical disease or psychiatric condition that, in the investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Time from commencement of treatment to disease progression or death, whichever occurs first, assessed up to 100 months
  To assess the progression free survival (PFS) for daratumumab in combination with thalidomide and dexamethasone in Asian patients with relapsed myeloma.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | anytime from commencement of treatment with daratumumab, thalidomide and dexamethasone to the end of studyaseline until disease progression, unmanageable adverse event or death, whichever occurs first, approximately up to 3 years
  percentage of patients enrolled that achieve a complete response (CR), or stringent complete response (sCR), or very good partial response (VGPR), or partial response (PR) based on the International Myeloma Working Group criteria
Overall survival (OS) | Up to approximately 5 years (anticipated) after the last participant is enrolled
  Time from commencement of treatment with daratumumab, thalidomide and dexamethasone to the date of death.
Duration of response (DOR) | the time from first evidence of PR or VGPR, or CR, or sCR to confirmation of disease progression or death due to any cause, assessed up to 100 months
  the time from first evidence of PR or VGPR, or CR, or sCR to confirmation of disease progression or death due to any cause.
Number of Participants affected by Adverse Events | from the time of enrolment into study till 3 years from the date of the last patient randomized
  assessed on the basis of the frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Wee Joo Chng, Principal Investigator — National University Hospital, Singapore
Locations (5):
- Queen Mary Hospital, Hong Kong, Hong Kong
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Samsung Medical Center, South Korea, South Korea
- National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Background] Lonial S, Weiss BM, Usmani SZ, Singhal S, Chari A, Bahlis NJ, Belch A, Krishnan A, Vescio RA, Mateos MV, Mazumder A, Orlowski RZ, Sutherland HJ, Blade J, Scott EC, Oriol A, Berdeja J, Gharibo M, Stevens DA, LeBlanc R, Sebag M, Callander N, Jakubowiak A, White D, de la Rubia J, Richardson PG, Lisby S, Feng H, Uhlar CM, Khan I, Ahmadi T, Voorhees PM. Daratumumab monotherapy in patients with treatment-refractory multiple myeloma (SIRIUS): an open-label, randomised, phase 2 trial. Lancet. 2016 Apr 9;387(10027):1551-1560. doi: 10.1016/S0140-6736(15)01120-4. Epub 2016 Jan 7. PMID 26778538
- [Background] Lokhorst HM, Plesner T, Laubach JP, Nahi H, Gimsing P, Hansson M, Minnema MC, Lassen U, Krejcik J, Palumbo A, van de Donk NW, Ahmadi T, Khan I, Uhlar CM, Wang J, Sasser AK, Losic N, Lisby S, Basse L, Brun N, Richardson PG. Targeting CD38 with Daratumumab Monotherapy in Multiple Myeloma. N Engl J Med. 2015 Sep 24;373(13):1207-19. doi: 10.1056/NEJMoa1506348. Epub 2015 Aug 26. PMID 26308596
- [Background] 3. Palumbo A, Chanan-Khan A, Weisel K, et al. Phase III randomized controlled study of daratumumab, bortezomib and dexamethasone (DVd) versus bortezomib and dexamethasone (Vd) in patients with relapsed or refractory multiple myeloma (RRMM): CASTOR study. J Clin Oncol 2016; 34 (Suppl abstr LBA4)
- [Background] 4. Dimopoulos MA, Oriol A, Nahi H, et al. An open-label, randomised phase 3 study of daratumumab, lenalidomide, dexamethasone (DRD) versus lenalidomide and dexamethasone (RD) in relapsed or refractory multiple myeloma (RRMM): POLLUX. EHA 2016 Abstract LB2238